CLINICAL TRIAL: NCT03521258
Title: Limb Salvage Through Tissue Engineering: A Novel Treatment Modality Using Dehydrated Human Amnion/Chorion Membrane
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Frank Lau, MD, Assistant Professor of Clinical Surgery, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9167
Record Dates: First submitted 2016-04-11; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Wounds; Trauma; Injury; Limb Salvage; Soft Tissue Injuries
MeSH Terms: conditions — Wounds and Injuries; Soft Tissue Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Human Amnion/Chorion Membrane + skin graft (Experimental): Dehydrated Human Amnion/Chorion Membrane (dHACM) will be placed on wound at the initial debridement to promote granulation tissue at the wound bed. Approximately 5-7 days following debridement, wound will be assessed for suitability of split thickness skin grafting. If an adequate granulation tissue is present, skin grafting will be performed and assessed for take in 5 days.
  Interventions: Device: Dehydrated Human Amnion/Chorion Membrane
- Flap Reconstruction (Standard of Care) (Active Comparator): A negative pressure wound dressing (NPWD) will be applied at the time of debridement until the wound is clean and adequate for flap reconstruction. Flap-based reconstruction is performed. Following flap reconstruction,patient will have 5 days of bed rest to allow proper healing and coverage of the wounds. If flaps are successful, patients starts a limb dangle protocol which gradually increases the dependent position and allows the flap to acclimate to new physiologic demands. Following dangle protocol patient will require inpatient physical and occupational therapy prior to discharge.
  Interventions: Procedure: Flap-Based Reconstructive Surgery

INTERVENTIONS:
Device: Dehydrated Human Amnion/Chorion Membrane
  Other Names: human amniotic membrane allograft; EpiFix
  Arms: Human Amnion/Chorion Membrane + skin graft
Procedure: Flap-Based Reconstructive Surgery — Standard of Care surgical intervention
  Arms: Flap Reconstruction (Standard of Care)

SUMMARY:
Extremity wounds with exposed critical structures, including bone and tendon are a major burden on the American healthcare system with limited treatment options. Free Flap reconstructions of lower extremity wounds have an increased failure rate in comparison to elective free flap procedures.These procedures are long and are associated with a high cost of care, prolonged hospital stays, and are limited by the need for surgical specialist availability and patient vessels suitable for anastomoses. This study will use a new treatment modality which is a commercially ready human amniotic membrane allograft (EpiFix) to promote a granulation tissue wound base that will be suitable for skin grafting, thus forgoing the need for a flap-based for reconstruction. The study goals are to reduce the overall cost of providing definitive treatment by decreasing operative time, length of hospital stay, decrease the need for intensive nursing care and rehabilitation. This study will aim to provide a treatment option that is readily accessible to all patients with these complex wounds in any healthcare setting across the country.

DETAILED DESCRIPTION:
53 patients ages 18 and over , presenting with wounds with exposed critical structures (bone and/or tendon) will be enrolled in the study and randomized into one of two groups. 21 patients will be in the standard treatment group (Flap based reconstruction) and 32 patients will be in the dHACM (EpiFix) + skin grafting treatment group (Experimental). Exclusion criteria includes exposed implanted hardware (surgical plates), anticipated need for future surgical procedures through the same wound, wounds resulting from surgical removal of malignancy, and patients who are not free flap candidates.

Data will be collected upon enrollment including:

Background and demographic information Wound size and severity Pain level Medication use Photographs of wound

Flap Reconstruction group (Standard of Care):

Patients in this group will have any dead, damaged or infected tissue removed from the wound and a negative pressure wound dressing will be applied until the wound is clean and adequate for flap reconstruction. Following flap reconstruction, patients typically require a 36-48 hour intensive care unit admission for flap monitoring and 5 days to bed rest to allow for proper healing. If the flap is successful, a dangle protocol will occur until patient increases the dependent position. Once the dangle protocol is completed, patients may require inpatient physical/occupational therapy prior to discharge from the hospital. If patient is not healing the physician may discuss other treatment options including crossing over to the EpiFix arm or amputation.

EpiFix and Skin Graft group:

Patients in this group will have any dead, damaged or infected tissue removed from wound. Once it is free from infection, a thin tissue (EpiFix) will be applied directly to the open wound. This will be covered by sterile wound dressing. After approximately 5-7 days the wound will be assessed for suitability of split thickness skin grafting. If adequately healed, skin grafting will be performed. After 5 days, the graft will be evaluated and if successful, the patient will be discharged home or to a rehab facility. If the wounds are not adequate for skin grafting, additional damaged tissue will removed and EpiFix will be placed until the wound is suitable for grafting. If you do not heal sufficiently the physician will discuss other treatment options including cross over to the standard of care Free Flap or amputation.

Study staff will evaluate the wound twice a week for the first 2 weeks, then once a week until 6 weeks. At this point, the patient will be followed every 4 weeks up to 22 weeks. Visits to the clinic will include wound measurements, photos, pain scale and evaluation of any infection.

ELIGIBILITY:
Inclusion Criteria:

* Wound includes exposed critical structures (tendon and/or bone)
* Patient is candidate flap reconstruction
* Patient is candidate for limb salvage

Exclusion Criteria:

* Wound involves weight-bearing surfaces (e.g. heel or forefoot wounds),
* Exposed implanted hardware (e.g. surgical plates)
* Anticipated need for future surgical procedures through the same wound
* Wounds resulting from surgical removal of malignancy
* Patients who are not flap candidates (e.g. severe peripheral vascular disease)
* Patients who are not limb salvage candidates (e.g. insensate or ischemic limbs).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | Within 6 weeks of treatment
  "Failure" will be defined as a composite of amputation, persistent exposed critical structures, development of osteomyelitis or need for additional flaps within 6 weeks of treatment.
  * Osteomyelitis will be diagnosed as pus from bone requiring long-term (>4 weeks) of IV antibiotics.),
  * Experimental Group: "Persistent exposed critical structures" in the experimental arm refers to persistence of exposed nerve, blood vessels, bone or tendon after 4 weeks of dHACM treatment
  * Standard of care group: Persistence of exposed nerve, blood vessels, bone or tendon after flap treatment

SECONDARY OUTCOMES:
Wound Issue | within 6 months of initial wound closure
  Were any of the following recorded: wound dehiscence, partial flap loss, or partial skin graft loss requiring prolonged local wound care or other wound treatment (e.g. hyperbaric oxygen therapy, negative pressure wound dressing, other wound devices)?
Epidermolysis | within 6 months of initial wound closure
  Was there any diagnosis of epidermolysis during study
Length of ICU stay | within 6 months of initial wound closure
  Total number of ICU inpatient days
Length of inpatient hospital stay | within 6 months of initial wound closure
  Total number of inpatient hospital days
Total treatment time from initial treatment to initial closure (excludes treatment of complications) | within 6 months of initial wound closure
  Total number of days from initial treatment to end of study
Total treatment time from initial treatment to completion of limb salvage (includes treatment of complications) | within 6 months of initial wound closure
  Total number of days from initial treatment to completion of limb salvage
Number of dHACM treatments required | within 6 months of initial wound closure
  Total number of EpiFix applications
Death from any cause | within 6 months of initial wound closure
  Death from any cause
Deep vein thrombosis diagnosed by radiologic imaging (e.g. ultrasound or CT) | within 6 months of initial wound closure
  Any diagnosis of DVT during study
Pulmonary embolus | within 6 months of initial wound closure
  Any diagnosis of PE during study
Ventilator-associated pneumonia | within 6 months of initial wound closure
  Any diagnosis of vent-associated pneumonia
Number of microsurgical revisions needed (arterial or venous) | within 6 months of initial wound closure
  Number of microsurgical revisions needed
Bony non union, bony melanin | within 6 months of initial wound closure
  Any diagnosis of bony non-union or bony melanin during study
Tendon rupture | within 6 months of initial wound closure
  Any diagnosis of tendon rupture during study

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lau, MD, Principal Investigator — Louisiana State University Health Sciences Center - New Orleans
Locations (1):
- Louisiana State University Health Sciences Center - N.O., New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kroll SS, Evans GR, Goldberg D, Wang BG, Reece GP, Miller MJ, Robb GL, Baldwin BJ, Schusterman MA. A comparison of resource costs for head and neck reconstruction with free and pectoralis major flaps. Plast Reconstr Surg. 1997 Apr;99(5):1282-6. doi: 10.1097/00006534-199704001-00011. PMID 9105354
- [Background] Hong S. Reconstructive surgery: lower extremity coverage. In: Plastic Surgery.Vol 4. 3rd ed. Elsevier Inc.; 2013:127-150.
- [Background] Colohan S, Saint-Cyr M. Management of lower extremity trauma. In: Plastic Surgery.Vol 4. 3rd ed. Elsevier Inc.; 2013:63-91.
- [Background] Chung KC, Saddawi-Konefka D, Haase SC, Kaul G. A cost-utility analysis of amputation versus salvage for Gustilo type IIIB and IIIC open tibial fractures. Plast Reconstr Surg. 2009 Dec;124(6):1965-1973. doi: 10.1097/PRS.0b013e3181bcf156. PMID 19952652
- [Background] MacKenzie EJ, Jones AS, Bosse MJ, Castillo RC, Pollak AN, Webb LX, Swiontkowski MF, Kellam JF, Smith DG, Sanders RW, Jones AL, Starr AJ, McAndrew MP, Patterson BM, Burgess AR. Health-care costs associated with amputation or reconstruction of a limb-threatening injury. J Bone Joint Surg Am. 2007 Aug;89(8):1685-92. doi: 10.2106/JBJS.F.01350. PMID 17671005
- [Background] Gore DC. Outcome and cost analysis for outpatient skin grafting. J Trauma. 1997 Oct;43(4):597-600; discussion 600-2. doi: 10.1097/00005373-199710000-00006. PMID 9356054
- [Background] Capla JM, Ceradini DJ, Tepper OM, Callaghan MJ, Bhatt KA, Galiano RD, Levine JP, Gurtner GC. Skin graft vascularization involves precisely regulated regression and replacement of endothelial cells through both angiogenesis and vasculogenesis. Plast Reconstr Surg. 2006 Mar;117(3):836-44. doi: 10.1097/01.prs.0000201459.91559.7f. PMID 16525274
- [Background] DeFranzo AJ, Argenta LC, Marks MW, Molnar JA, David LR, Webb LX, Ward WG, Teasdall RG. The use of vacuum-assisted closure therapy for the treatment of lower-extremity wounds with exposed bone. Plast Reconstr Surg. 2001 Oct;108(5):1184-91. doi: 10.1097/00006534-200110000-00013. PMID 11604617
- [Background] Hovius SER, Kan HJ, Smit X, Selles RW, Cardoso E, Khouri RK. Extensive percutaneous aponeurotomy and lipografting: a new treatment for Dupuytren disease. Plast Reconstr Surg. 2011 Jul;128(1):221-228. doi: 10.1097/PRS.0b013e31821741ba. PMID 21701337
- [Background] Godina M. Early microsurgical reconstruction of complex trauma of the extremities. Plast Reconstr Surg. 1986 Sep;78(3):285-92. doi: 10.1097/00006534-198609000-00001. PMID 3737751
- [Background] Parrett BM, Matros E, Pribaz JJ, Orgill DP. Lower extremity trauma: trends in the management of soft-tissue reconstruction of open tibia-fibula fractures. Plast Reconstr Surg. 2006 Apr;117(4):1315-22; discussion 1323-4. doi: 10.1097/01.prs.0000204959.18136.36. PMID 16582806
- [Background] Khouri RK, Cooley BC, Kunselman AR, Landis JR, Yeramian P, Ingram D, Natarajan N, Benes CO, Wallemark C. A prospective study of microvascular free-flap surgery and outcome. Plast Reconstr Surg. 1998 Sep;102(3):711-21. doi: 10.1097/00006534-199809030-00015. PMID 9727436
- [Background] Stern M. THE GRAFTING OF PRESERVED AMNIOTIC MEMBRANE TO BURNED AND ULCERATED SURFACES, SUBSTITUING SKIN GRAFTS. JAMA. 1913;60(13):973-974.
- [Background] Gruss JS, Jirsch DW. Human amniotic membrane: a versatile wound dressing. Can Med Assoc J. 1978 May 20;118(10):1237-46. PMID 647542
- [Background] Zelen CM, Gould L, Serena TE, Carter MJ, Keller J, Li WW. A prospective, randomised, controlled, multi-centre comparative effectiveness study of healing using dehydrated human amnion/chorion membrane allograft, bioengineered skin substitute or standard of care for treatment of chronic lower extremity diabetic ulcers. Int Wound J. 2015 Dec;12(6):724-32. doi: 10.1111/iwj.12395. Epub 2014 Nov 26. PMID 25424146
- [Background] Sheikh ES, Sheikh ES, Fetterolf DE. Use of dehydrated human amniotic membrane allografts to promote healing in patients with refractory non healing wounds. Int Wound J. 2014 Dec;11(6):711-7. doi: 10.1111/iwj.12035. Epub 2013 Feb 15. PMID 23409746
- [Background] Serena TE, Carter MJ, Le LT, Sabo MJ, DiMarco DT; EpiFix VLU Study Group. A multicenter, randomized, controlled clinical trial evaluating the use of dehydrated human amnion/chorion membrane allografts and multilayer compression therapy vs. multilayer compression therapy alone in the treatment of venous leg ulcers. Wound Repair Regen. 2014 Nov-Dec;22(6):688-93. doi: 10.1111/wrr.12227. Epub 2015 Jan 8. PMID 25224019
- [Background] Siegel JE, Weinstein MC, Russell LB, Gold MR. Recommendations for reporting cost-effectiveness analyses. Panel on Cost-Effectiveness in Health and Medicine. JAMA. 1996 Oct 23-30;276(16):1339-41. doi: 10.1001/jama.276.16.1339. PMID 8861994
- [Background] Koob TJ, Rennert R, Zabek N, Massee M, Lim JJ, Temenoff JS, Li WW, Gurtner G. Biological properties of dehydrated human amnion/chorion composite graft: implications for chronic wound healing. Int Wound J. 2013 Oct;10(5):493-500. doi: 10.1111/iwj.12140. Epub 2013 Aug 1. PMID 23902526
- [Background] Robson MC, Krizek TJ. The effect of human amniotic membranes on the bacteria population of infected rat burns. Ann Surg. 1973 Feb;177(2):144-9. doi: 10.1097/00000658-197302000-00003. No abstract available. PMID 4633388
- [Derived] Lau FH, Hoffman RD, Danos D, Torabi R, Patterson CW, McKendrick AD, Stalder M, Dupin C, Hilaire HS. Regenerative vs flap-based limb salvage: a multi-centered, prospective, randomized controlled trial. Regen Med. 2023 Mar;18(3):207-218. doi: 10.2217/rme-2022-0147. Epub 2023 Feb 16. PMID 36794542